CLINICAL TRIAL: NCT05755932
Title: A Randomized, Double-blind, Two-way Crossover Study to Assess the Effect of Hydrofluoroolefin (HFO) Propellant Metered Dose Inhaler (MDI) on Mucociliary Clearance Compared With Hydrofluoroalkane (HFA) Propellant MDI in Healthy Participants
Brief Title: Study to Assess Effect of Next-Generation Propellant MDI on Mucociliary Clearance Vs. HFA Propellant MDI in Healthy Participants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: D5985C00006
Record Dates: First submitted 2023-02-23; First posted 2023-03-06 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Mucociliary Clearance
Keywords: Mucociliary Clearance, Propellant
MeSH Terms: interventions — norflurane

STUDY DESIGN:
Intervention Model Description: A randomized, double-blind, multi-site, two-way crossover study to assess the effect on MCC and safety of HFO propellant compared to HFA propellant in healthy participants. Mucociliary clearance will be determined after 1 week of twice daily (BID) administration of HFO MDI (test) and HFA MDI (reference). Study treatment will be administered via MDI device as 6 inhalations BID Participants will receive treatments in 1 of 2 possible treatment sequences: A followed by B, or B followed by A.
  * Treatment A: HFO MDI - test formulation
  * Treatment B: HFA MDI - reference formulation The study will comprise
  * A Screening Period 7 to 14 days prior to first dosing;
  * Two Treatment Periods (TPs) of 7 days each, a 7 to 14 day Washout Period between the 2 TPs; and
  * A final safety Follow-up Visit
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study is double blinded with regard to treatment (MDI administered with 2 different propellants [Treatment A or B]), ie, the sponsor, the investigator, all clinical staff involved in the clinical study, the participants, and the study monitor will remain blinded, unless safety concerns or a regulatory requirement necessitate unblinding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment A: HFO MDI (Experimental): Test arm, 6 inhalations BID for 7 days
  Interventions: Drug: HFO-1234ze(E)
- Treatment B: HFA MDI (Active Comparator): Reference arm, 6 inhalations BID for 7 days
  Interventions: Drug: HFA-134a

INTERVENTIONS:
Drug: HFO-1234ze(E) — * Dose formulation: metered dose inhaler (MDI)
  * Unit dose strength(s): Experimental (propellant only)
  * Dosage level(s): 6 inhalations, BID
  * Route of administration: Oral inhalation
  * Participants will receive treatment A in 1 of 2 possible treatment sequences: AB or BA
  Other Names: Propellant in MDI
  Arms: Treatment A: HFO MDI
Drug: HFA-134a — * Dose formulation: metered dose inhaler (MDI)
  * Unit dose strength(s): Reference (propellant only)
  * Dosage level(s): 6 inhalations, BID
  * Route of administration: Oral inhalation
  * Participants will receive treatment B in 1 of 2 possible treatment sequences: AB or BA.
  Other Names: Propellant in MDI
  Arms: Treatment B: HFA MDI

SUMMARY:
A Study to Assess the Effect of the HFO MDI Propellant on Mucociliary Clearance Compared to the HFA MDI Propellant in Healthy Participants

DETAILED DESCRIPTION:
A randomized, double-blind, multi-site, two-way crossover study to assess the effect on MCC and safety of HFO propellant compared to HFA propellant in healthy participants. Mucociliary clearance will be determined after 1 week of twice daily (BID) administration of HFO MDI (test) and HFA MDI (reference).

The study will comprise a Screening Period 7 to 14 days prior to first dosing; Two Treatment Periods (TPs) of 7 days each (+ up to 3 days), with a 7 to 14 day Washout Period between the 2 TPs; and a final safety Follow-up Visit 5 to 7 days after the final dose administration in TP2.

Participants will receive treatments in 1 of 2 possible treatment sequences: A followed by B, or B followed by A.

Study treatment will be administered via MDI device as 6 inhalations BID (every morning and evening approximately 12 hours apart):

Treatment A: HFO MDI; 6 inhalations per dose - test formulation Treatment B: HFA MDI; 6 inhalations per dose - reference formulation

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible to be included in the study only if all of the following criteria apply:

1. Capable of giving signed informed consent as described in the protocol which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.
2. Healthy non-smoking male and/or female participants aged 18 to 60 years inclusive at the time of signing the informed consent, without respiratory comorbidities.
3. Participant must have a forced expiratory volume in 1 second (FEV1) ≥ 80% of the predicted value for age, height, and ethnicity at screening, and FEV1/forced vital capacity (FVC) ratio of > 70%.
4. Participant must demonstrate acceptable MDI administration using empty training MDI.
5. Participant willing to comply with study IP administration requirements, defined as ≥ 80% participant medication adherence during the Treatment Periods.
6. Body mass index (BMI) within the range 18 to 35 kg/m2 (inclusive), and weight within the range 50 to 120 kg (inclusive).
7. Female participants must be not of childbearing potential or must use a form of highly effective birth control as defined below:

   (a) Women not of childbearing potential are defined as women who are either permanently sterilized (hysterectomy, bilateral oophorectomy, or bilateral salpingectomy), or who are postmenopausal. Women will be considered postmenopausal if they have been amenorrheic for 12 months prior to the planned date of randomization without an alternative medical cause. The following age-specific requirements apply:
   * Women < 50 years old would be considered postmenopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatment and follicle stimulating hormone (FSH) levels in the postmenopausal range.
   * Women ≥ 50 years old would be considered postmenopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatment.
8. Female participants of childbearing potential must use one highly effective form of birth control. A highly effective method of contraception is defined as one that can achieve a failure rate of less than 1% per year when used consistently and correctly. At enrollment, women of childbearing potential who are sexually active with a non-sterilized male partner should be stable on their chosen method of highly effective birth control, as defined below, and willing to remain on the birth control until at least 14 days after last dose of study intervention. Cessation of contraception after this point should be discussed with a responsible physician. Periodic abstinence (calendar, symptothermal, post-ovulation methods), withdrawal (coitus interruptus), spermicides only, and lactational amenorrhea method are not acceptable methods of contraception. Female condom and male condom should not be used together.

   * All women of childbearing potential must have a negative serum pregnancy test result at Visit 1.

     * Females <50 years of age with amenorrhea for 12 months without an alternative medical cause must have a serum FSH test at Visit 1.
     * Highly effective birth control methods are listed below:
   * Total sexual abstinence is an acceptable method provided it is the usual lifestyle of the participant (defined as refraining from heterosexual intercourse during the entire period of risk associated with the study treatments).
   * Combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation:

     * Oral
     * Intravaginal
     * Transdermal
   * Progestogen-only hormonal contraception associated with inhibition of ovulation:

     * Oral
     * Injectable
     * Implantable
   * Intrauterine device or intrauterine hormone-releasing system
   * Bilateral tubal occlusion
   * Male partner sterilization/vasectomy with documentation of azoospermia prior to the female participant's entry into the study, and this male is the sole partner for that participant. The documentation on male sterility can come from the site personnel's review of participant's medical records, medical examination and/or semen analysis or medical history interview provided by her or her partner.

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

1. History of smoking > 10 pack-years, or participant quit smoking < 6 months prior to screening.
2. Acute or chronic upper or lower respiratory illness within 30 days of screening.
3. Respiratory medication or medication impacting ciliary clearance for any indication within 30 days of screening.
4. History of more than 2 chest CTs or equivalent (> 10 mSv) within the past year.
5. History of any clinically significant disease or disorder which, in the opinion of the investigator, may either put the participant at risk because of participation in the study, or influence the results or the participant's ability to participate in the study.
6. Any clinically significant illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of the IP.
7. History of any cancer except squamous cell and basal cell carcinomas of the skin.
8. Any clinically significant abnormalities in clinical chemistry, hematology, or urinalysis results, at screening as judged by the investigator.
9. Any clinically significant abnormal findings in vital signs at screening, as judged by the investigator.
10. Any clinically significant abnormalities on 12-lead ECG at screening, as judged by the investigator. Note: Participants with ECG QT interval corrected for heart rate using Fridericia's formula (QTcF) > 480 msec will be excluded.
11. A SARS-CoV-2 infection in the 8 weeks prior to Visit 1, or during the Screening Period, or that required hospitalization at any time prior to Visit 1 or during the Screening Period.
12. Participant has clinical signs and symptoms consistent with SARS-CoV-2 infection; eg, fever, dry cough, dyspnea, sore throat, fatigue, or laboratory-confirmed acute infection with SARS-CoV-2.
13. Participant who had severe course of COVID-19 (extracorporeal membrane oxygenation, mechanically ventilated, Intensive Care Unit stay).
14. History of any respiratory disorders such as asthma, chronic obstructive pulmonary disease, or idiopathic pulmonary fibrosis, alpha-1 antitrypsin, primary ciliary dyskinesia, cystic fibrosis.
15. Known or suspected history of drug abuse, as judged by the investigator.
16. Current smokers or those who have smoked or used nicotine products (including electronic cigarettes) marijuana, vaping, etc, within the 6 months prior to screening.
17. Positive screen for drugs of abuse or cotinine at screening.
18. Use of any prescribed or non-prescribed medication including antacids, analgesics (other than paracetamol/acetaminophen), herbal remedies, megadose of vitamins (intake of 20 to 600 times the recommended daily dose), and minerals within 14 days or 5 half-lives (whichever is longer) prior to the first administration of IP.
19. Excessive intake of caffeine-containing drinks or food (eg, coffee, tea, chocolate) as judged by the investigator. Excessive intake of caffeine defined as the regular consumption of more than 600 mg of caffeine per day (eg, > 5 cups of coffee) or would likely be unable to refrain from the use of caffeine-containing beverages.
20. Using any herbal products either by inhalation or by nebulizer within 2 weeks of Visit 1, and does not agree to stop for the duration of the study.
21. Participation in another clinical study with an IP administered in the last 30 days or 5 half-lives, whichever is longer.
22. Involvement of any AstraZeneca, Fortrea, or study site employee or their close relatives.
23. Participants who have previously received HFO via inhalation (eg, BGF [also known as PT010, Breztri, Trixeo] HFO).
24. Judgment by the investigator that the participant should not participate in the study if they have any ongoing or recent (ie, during the Screening Period) minor medical complaints that may interfere with the interpretation of study data or are considered unlikely to comply with study procedures, restrictions, and requirements.
25. Participants who cannot communicate reliably with the investigator.
26. Vulnerable participants, eg, kept in detention, protected adults under guardianship, trusteeship, or committed to an institution by governmental or judicial order.
27. Female participants who are currently pregnant (confirmed with positive pregnancy test), breast feeding, or planned pregnancy during the study or women of childbearing potential not using acceptable contraception measures (see Inclusion Criterion).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2023-06-14 (Actual); Primary Completion 2024-07-22 (Actual); Study Completion 2024-07-22 (Actual)

PRIMARY OUTCOMES:
Change from baseline in MCC through 60 minutes following inhalation of 99m technetium-labelled colloid (sulfur or albumin) colloid and gamma camera imaging. | 7 days
  Change from baseline in MCC through 60 minutes, following inhalation of 99m technetium-labelled colloid (sulfur or albumin) and gamma camera imaging

SECONDARY OUTCOMES:
Change from baseline in MCC at 3 hours following inhalation of 99m technetium-labelled colloid (sulfur or albumin)and gamma camera imaging | 7 days
  Change from baseline in MCC at 3 hours, following inhalation of 99m technetium-labelled colloid (sulfur or albumin) and gamma camera imaging

OTHER OUTCOMES:
Safety and tolerability will be evaluated in terms of AEs | up to 35 days
  To assess the safety and tolerability after administration of HFO MDI as compared to HFA MDI in healthy participants

CONTACTS AND LOCATIONS:
Overall Officials: William D Bennett, PhD, Principal Investigator — University of North Carolina, Chapel Hill; Andreas Schmid, MD, Principal Investigator — University of Kansas Medical Center; Timothy Corcoran, PhD, Principal Investigator — UPMC Montefiore Hospital; Peter Mogayzel, MD, PhD, MBA, Principal Investigator — Johns Hopkins University; Douglas Conrad, MD, Principal Investigator — University of California, San Diego
Locations (5):
- United States (4):
  - Research Site, Kansas City, Kansas
  - Research Site, Baltimore, Maryland
  - Research Site, Chapel Hill, North Carolina
  - Research Site, Pittsburgh, Pennsylvania
- Research Site, Glasgow, United Kingdom

REFERENCES:
- [Result] Graham BL, Steenbruggen I, Miller MR, Barjaktarevic IZ, Cooper BG, Hall GL, Hallstrand TS, Kaminsky DA, McCarthy K, McCormack MC, Oropez CE, Rosenfeld M, Stanojevic S, Swanney MP, Thompson BR. Standardization of Spirometry 2019 Update. An Official American Thoracic Society and European Respiratory Society Technical Statement. Am J Respir Crit Care Med. 2019 Oct 15;200(8):e70-e88. doi: 10.1164/rccm.201908-1590ST. PMID 31613151
- [Result] Investigator's Brochure - Budesonide, Glycopyrronium and Formoterol Fumarate Inhalation Aerosol (BGF MDI); Budesonide and Formoterol Fumarate Inhalation Aerosol (BFF MDI); Budesonide Inhalation Aerosol (BD MDI); Glycopyrronium Inhalation Aerosol (GP MDI) (Also known as PT010 [BGF MDI], PT009 [BFF MDI], PT008 (BD MDI); PT001 (GP MDI); Edition Number 8.0, 22 April 2020.
- [Result] Quanjer PH, Stanojevic S, Cole TJ, Baur X, Hall GL, Culver BH, Enright PL, Hankinson JL, Ip MS, Zheng J, Stocks J; ERS Global Lung Function Initiative. Multi-ethnic reference values for spirometry for the 3-95-yr age range: the global lung function 2012 equations. Eur Respir J. 2012 Dec;40(6):1324-43. doi: 10.1183/09031936.00080312. Epub 2012 Jun 27. PMID 22743675
- [Result] Laube BL, Carson KA, Sharpless G, Paulin LM, Hansel NN. Mucociliary Clearance in Former Tobacco Smokers with Both Chronic Obstructive Pulmonary Disease and Chronic Bronchitis and the Effect of Roflumilast. J Aerosol Med Pulm Drug Deliv. 2019 Aug;32(4):189-199. doi: 10.1089/jamp.2018.1459. Epub 2019 Apr 8. PMID 30964381
- [Result] Bennett WD, Wu J, Fuller F, Balcazar JR, Zeman KL, Duckworth H, Donn KH, O'Riordan TG, Boucher RC, Donaldson SH. Duration of action of hypertonic saline on mucociliary clearance in the normal lung. J Appl Physiol (1985). 2015 Jun 15;118(12):1483-90. doi: 10.1152/japplphysiol.00404.2014. Epub 2015 Apr 24. PMID 25911685